CLINICAL TRIAL: NCT01181271
Title: Sequential Myeloablative Autologous Stem Cell Transplantation Followed by Allogeneic Non-Myeloablative Stem Cell Transplantation for Patients With Poor Risk Lymphomas
Brief Title: Tandem Auto-Allo Transplant for Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-057
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Diffuse, Large B-Cell, Lymphoma; Lymphoma, Low-Grade; T-Cell Lymphoma; Mantle-Cell Lymphoma; Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Lymphoma, Small Lymphocytic
Keywords: Lymphoma; non-hodgkins lymphoma; Hodgkin's lymphoma; Hodgkin's disease; stem cell transplant; High-risk diffuse large B cell; Transformed low grade lymphoma; T-cell non-Hodgkin's lymphoma; Mantle cell lymphoma at any time in therapy; "Double-hit" lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Lymphoma, Mantle-Cell; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — Busulfan; Etoposide; Cyclophosphamide; Mesna; Peripheral Blood Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; fludarabine phosphate; Transplantation; Tacrolimus; Sirolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous then Allogeneic transplant (Experimental): All patients will receive conditioning with busulfan, etoposide, and cyclophosphamide (with mesna) and then will undergo autologous (auto) peripheral blood stem cell transplantation.
  Patients will be re-evaluated after autologous transplant prior to proceeding to non-myeloablative allogeneic (allo) transplant. If eligible to proceed, allogenic transplantation will take place no earlier than 40 days and no later than 180 days after autologous stem cell transplantation.
  Conditioning for the allogeneic transplant will consist of fludarabine and busulfan. Participants will receive tacrolimus and sirolimus as prophylaxis against graft versus host disease (GVHD).
  Interventions: Drug: Busulfan (conditioning for AUTO transplant); Drug: Etoposide (conditioning for AUTO transplant); Drug: Cyclophosphamide (conditioning for AUTO transplant); Drug: Mesna (prior to AUTO transplant); Other: autologous (auto) peripheral blood stem cell transplantation; Drug: Neupogen; Drug: Fludarabine (conditioning for ALLO Transplant); Drug: Busulfan (conditioning for ALLO Transplant); Other: non-myeloablative allogeneic (allo) transplant; Drug: Tacrolimus; Drug: Sirolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Busulfan (conditioning for AUTO transplant) — 0.8 mg/kg intravenous (IV) bolus every six hours (Q6H) on days -8,-7,-6,-5 (total of 14 doses). The total daily dose of busulfan will be 3.2 mg/kg on days -8,-7, and -6 and 1.6 mg/kg on day -5
  Other Names: Busulfex
Drug: Etoposide (conditioning for AUTO transplant) — Etoposide 30 mg/kg IV bolus every day (QD) on day -4. The total daily dose of etoposide will be 30 mg/kg.
  Other Names: VP-16
Drug: Cyclophosphamide (conditioning for AUTO transplant) — Cyclophosphamide 60 mg/kg IV bolus QD on days -3 and -2. The total daily dose of cyclophosphamide will be 60 mg/kg.
  Other Names: Cytoxan
Drug: Mesna (prior to AUTO transplant) — Mesna 15 mg/kg IV bolus on days -3 and -2 infused over 15 minutes and given 15 minutes prior to cyclophosphamide administration. This is followed by Mesna given 15 mg/kg IV bolus three times daily (TID) on days -3 and -2 infused over 15 minutes at 3, 6, and 9 hours after completion of cyclophosphamide infusion. Total daily dose of Mesna should be equivalent to daily dose of cyclophosphamide. Lastly, Mesna will be given at 15 mg/kg IV bolus QD on day -1. This makes a total of 9 doses of Mesna
Other: autologous (auto) peripheral blood stem cell transplantation — Infusion of autologous peripheral blood stem cells on Day 0.
Drug: Neupogen — Neupogen 5 mcg/kg subcutaneous (SQ) daily starting on day +1 until absolute neutrophil count (ANC) is greater than or equal to 1000 per micro liter on two separate occasions or greater than 5000 per micro liter once
  Other Names: G-CSF
Drug: Fludarabine (conditioning for ALLO Transplant) — Fludarabine 30 mg/m2/day will be administered as a bolus infusion over approximately 30 minutes for 4 days on days -5, -4, -3, -2.
  Other Names: Fludara
Drug: Busulfan (conditioning for ALLO Transplant) — Busulfan will be administered by IV infusion over approximately 3 hours on days -5, -4, -3, -2. The dose of busulfan will be 0.8 mg/kg/day
  Other Names: Busulfex
Other: non-myeloablative allogeneic (allo) transplant — Donor peripheral blood stem cells (PBSC) will be infused intravenously beginning on Day 0. The minimum total CD34+ cell dose will be 2 x 10^6 CD34+cells/kg of recipient's actual body weight with a maximum dose of 8 x 10^6/kg of recipient's actual body weight
Drug: Tacrolimus — Tacrolimus (FK506) will be given orally at a dose of 0.05 mg/kg orally (PO) twice a day (BID) starting day -3.
  Other Names: FK506
Drug: Sirolimus — Sirolimus (rapamycin) will be given orally at a dose of 12 mg times one on day -3 and then the dose shall be 4 mg by mouth daily starting on day -2. The dose may then be adjusted according to serum levels at the discretion of the treating physician
  Other Names: Rapamycin
Drug: Methotrexate — Methotrexate will be administered once daily on days 1, 3, and 6 as an IV bolus over 15 minutes at a dose of 5 mg/m2

SUMMARY:
Relapse remains a principle cause of treatment failure for patients with aggressive lymphoma after autologous transplantation. Non-myeloablative allogeneic transplantation allows patients to receive an infusion of donor cells in an attempt to induce a graft versus lymphoma effect. This study will assess the feasibility, safety and efficacy of the combination of autologous stem cell transplantation followed by non-myeloablative transplantation for patients with poor-risk aggressive lymphoma.

DETAILED DESCRIPTION:
This is a phase II clinical trial investigating the feasibility, and efficacy of sequential autologous stem cell transplant followed by non-myeloablative allogeneic transplant for patients with poor risk lymphoma. Patients will be enrolled onto the trial when eligible and undergo standard high-dose chemotherapy with the combination with busulfan, cyclophosphamide, and etoposide followed by autologous stem cell transplant. After recovery of counts and clinical status, patients will then proceed to non-myeloablative allogeneic stem cell transplant using a fully matched related or unrelated donor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk diffuse large B cell or transformed low grade lymphoma defined as:

  * Residual disease after at least 6 cycles of anthracycline-based chemotherapy (with residual disease defined as persistent bone marrow involvement and/or persistent measurable lymph node or solid organ masses that are PET or gallium avid)
  * Progressive disease after at least 2 cycles of anthracycline-based chemotherapy
  * Patients with an initial complete response but subsequent relapse within 6 months after completion of anthracycline-based chemotherapy
* Patients with any T-cell non-Hodgkin's lymphoma as defined as:

  * Peripheral T-cell lymphoma (ALK negative PTCL-U) including PTCL-NOS, HSGD (hepato-splenic gamma-delta TCL), AITL (angioimmunoblastic T-cell lymphoma), EATL (enteropathy associated T-cell lymphoma), ALK-negative anaplastic large cell lymphoma
  * Any T-cell histology (except LGL) with residual disease after at least 4 cycles of anthracycline-based chemotherapy (with residual disease defined as persistent bone marrow involvement and/or persistent measurable lymph node or solid organ masses that are PET or gallium avid)
* Patients with mantle cell lymphoma at any time in therapy
* Patients with "double-hit" lymphoma as characterized by the presence of concurrent overexpression of Bcl-2 and c-myc
* Patients with Hodgkin's lymphoma that is

  * Refractory to first-line therapy and at least one second line chemotherapy regimen
  * Relapsed Hodgkin's lymphoma which is refractory to at least one salvage chemotherapy regimen.
* Patients with CLL/SLL with 17p- cytogenetic abnormality
* Age 18 years and greater
* ECOG performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document.
* Responsive disease to last therapy as determined by at least one of the following:

  * At least PR by Revised Response Criteria
  * At least PR by traditional Cheson Criteria
  * < 10% of overall cellularity involved with disease on bone marrow biopsy for patients with involvement of the bone marrow
* Minimum of 2 x 106 CD34+ cells / kg already collected and frozen. These stem cells may have been collected from PBSC pheresis, bone marrow harvest, or the combination.

Exclusion Criteria:

Patients will be re-evaluated after autologous transplant prior to proceeding to non-myeloablative transplant

* Pregnancy
* Evidence of HIV infection
* Heart failure uncontrolled by medications or ejection fraction less than 45%
* Active involvement of the CNS by lymphoma
* Inability to provide informed consent
* Previous autologous or allogeneic stem cell transplant
* Creatinine greater than 2 gm/dL or 24 hour urine creatinine clearance < 50 cc/minute (does not have to satisfy both)
* Total bilirubin greater than 2 times the upper limit of normal except when due to Gilbert's syndrome or hemolysis.
* Transaminases greater than 3 times the upper limit of normal
* FVC or DLCO of less than 50% of predicted (DLCO corrected for hemoglobin level)
* Already known to not possess suitably HLA-matched related or unrelated donor

Eligibility to proceed to allogeneic transplant Cannot be admitted for allogeneic transplant earlier than 40 days and no later than 180 days after autologous stem cell transplant.

* HLA identical (A, B, C and DR) related or unrelated donor available. HLA typing of class I loci (HLA- A, B, C) will be based on complement dependent cytotoxicity assay or PCR of sequence specific oligonucleotide primers (SSOP). Typing of HLA class II (DRB1) will be based on PCR of sequence specific oligonucleotide primers (SSOP).
* No need for intravenous hydration in the previous 2 weeks
* Resolved mucositis
* Renal, cardiac, pulmonary, and hepatic function meet standard criteria for nonmyeloablative SCT as listed below:

  * Serum Cr < 2 gm/dL
  * LV ejection fraction > 30% and no uncontrolled symptoms of congestive heart failure
  * DLCO > 50% of predicted value (corrected for hemoglobin)
  * Transaminases < 5X the institution upper limit of normal
  * Bilirubin < 3X the institution upper limit of normal except when Gilbert's Syndrome or hemolysis is present
  * ECOG PS ≤ 2
* No intravenous antimicrobials within 2 weeks
* No evidence of progressive disease, defined as a 25% increase from nadir in the sum of the product of the diameters (SPD) of any lymph node previously identified as abnormal prior to autologous transplant or the appearance of any new lymph node greater than 1.5 cm in greatest diameter, new bone marrow involvement, or new solid organ nodule greater than 1 cm in diameter. This restaging study will be performed at least 28 days after the autologous transplant and within 60 days prior to admission for allogeneic transplant. Status of stable disease (SD) is acceptable to proceed to allogeneic transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin A Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen YB, Li S, Fisher DC, Driscoll J, Del Rio C, Abramson J, Armand P, Barnes J, Brown J, Cutler C, El-Jawahri A, Ho VT, Hochberg E, McAfee S, Takvorian R, Spitzer TR, Antin JH, Soiffer R, Jacobsen E. Phase II Trial of Tandem High-Dose Chemotherapy with Autologous Stem Cell Transplantation Followed by Reduced-Intensity Allogeneic Stem Cell Transplantation for Patients with High-Risk Lymphoma. Biol Blood Marrow Transplant. 2015 Sep;21(9):1583-8. doi: 10.1016/j.bbmt.2015.05.016. Epub 2015 May 22. PMID 26009261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between October 2010 and June 2013.
Groups:
- Autologous Then Allogeneic Transplant: Autologous, then Allogeneic Stem Cell Transplantation
Period: Autologous Transplant
Arm/Group | Autologous Then Allogeneic Transplant
Started | 42
Completed | 42
Not Completed | 0
Period: Evaluation for Allogeneic Transplant
Arm/Group | Autologous Then Allogeneic Transplant
Started | 42
Completed | 29
Not Completed | 13
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 4
Not completed — No suitable donor | 2
Not completed — therapy-related AML diagnosed | 1
Period: Allogeneic Transplant
Arm/Group | Autologous Then Allogeneic Transplant
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Autologous Then Allogeneic Transplant: Autologous then allogeneic stem cell transplantation
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 56.5 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Prior lines of chemotherapy [Median (Full Range); unit: lines] | 2 [1 to 6]
Diagnosis [Count of Participants; unit: Participants]
  Relapsed/refractory Diffuse Large B-cell Lymphoma | 10
  Relapsed/refractory Non-Hodgkin Lymphoma | 6
  Double-Expressing Non-Hodgkin Lymphoma | 9
  Transformed B-cell Non-Hodgkin Lymphoma | 8
  T-cell Non-Hodgkin Lymphoma | 4
  Mantle cell Non-Hodgkin Lymphoma | 3
  Relapsed/Refractory Hodgkin Lymphoma | 1
  Heavy chain disease | 1
Disease status at study entry [Count of Participants; unit: Participants]
  Partial Response | 21
  Complete Response | 21

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Blood All-cell Donor Chimerism
Description: Successful donor stem cell engraftment is defined as when ≥ 80% of hematopoietic elements are donor-derived as determined by chimerism assays from peripheral blood at day 100 after non-myeloablative allogeneic stem cell transplantation.
Time Frame: 100 days post allogeneic transplant
Population: Participants who underwent the full tandem AUTO-ALLO stem cell transplant
Measure: Median (Full Range); unit: percentage of donor-derived elements
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of donor-derived elements | 95 [83 to 99]

2. Secondary Outcome: Number of Days After Allogeneic Transplant Until Absolute Neutrophil Count Was Equal to or Greater Than 500/uL
Time Frame: within 28 days after allogeneic transplant
Population: This was only measured in the 17 participants who experienced a hematological nadir after allo transplant.
Measure: Median (Full Range); unit: days
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 17
days | 12 [1 to 18]

3. Secondary Outcome: Cumulative Incidence of Grades II to IV Acute Graft Versus Host Disease (GVHD)
Description: Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: within 200 days after allogeneic transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of participants | 13.8 [5.3 to 26.3]

4. Secondary Outcome: Cumulative Incidence of Extensive Chronic Graft-versus-host-disease
Description: Extensive chronic graft versus-host-disease (GVHD) was defined as GVHD that required systemic immunosuppression.
Time Frame: 1-year after allogeneic transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of participants | 37.9 [23.1 to 52.7]

5. Secondary Outcome: Cumulative Incidence of Non-relapse Mortality
Description: Non-relapse mortality is defined as participants who die from causes other than their underlying disease relapse, such as infection or graft versus host disease
Time Frame: 2-years after allogeneic transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of participants | 11.1 [3.5 to 23.6]

6. Secondary Outcome: Cumulative Incidence of Disease Relapse
Time Frame: 2-years after allogeneic transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of participants | 17.2 [7.5 to 30.4]

7. Secondary Outcome: Estimated Two Year Progression Free Survival Rate for Participants Undergoing Both Autologous and Allogeneic Transplants
Time Frame: 2 years after allogeneic transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of participants | 72 [55 to 83]

8. Secondary Outcome: Estimated Two Year Overall Survival Rate for Participants Undergoing Both Autologous and Allogeneic Transplants
Time Frame: Two-years after Allogeneic Transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 29
percentage of participants | 89 [74 to 96]

9. Secondary Outcome: Estimated Two Year Progression Free Survival Rate for All Participants
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 42
percentage of participants | 64 [50 to 75]

10. Secondary Outcome: Estimated Two Year Overall Survival Rate for All Participants
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 42
percentage of participants | 83 [70 to 90]

11. Secondary Outcome: Estimated Two Year Progression Free Survival Rate for Participants Undergoing Only Autologous Transplant
Time Frame: Two Years
Population: Participants who ONLY underwent Autologous transplant (did not proceed to Allogeneic)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 13
percentage of participants | 46 [23 to 66]

12. Secondary Outcome: Estimated Two Year Overall Survival Rate for Participants Undergoing Only Autologous Transplant
Time Frame: two years
Population: Participants who ONLY underwent Autologous transplant, did not proceed to Allogeneic transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Then Allogeneic Transplant
Number analyzed (Participants) | 13
percentage of participants | 69 [43 to 85]

ADVERSE EVENTS:
Time Frame: Until 30 months after allogeneic transplant.
Arm/Group | Autologous Then Allogeneic Transplant
Serious Adverse Events (participants affected / at risk) | 5/42
Other Adverse Events (participants affected / at risk) | 24/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous Then Allogeneic Transplant (N=42)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
sepsis (Infections and infestations) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Death, not otherwise specified (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous Then Allogeneic Transplant (N=42)
anemia (Blood and lymphatic system disorders) | 4
febrile neutropenia (Blood and lymphatic system disorders) | 5
colitis (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 4
mucositis oral (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 3
edema (General disorders) | 2
neutrophil count decreased (Investigations) | 2
platelet count decreased (Investigations) | 6
weight loss (Investigations) | 2
muscle weakness (Musculoskeletal and connective tissue disorders) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes